CLINICAL TRIAL: NCT07251439
Title: Impact of Perioperative Body Temperature on Postoperative Complications and Pain in Video-assisted Thoracoscopic Surgery Patients Utilizing Continuous Temperature Monitoring: A Prospective Cohort Study
Brief Title: Impact of Perioperative Body Temperature on Postoperative Complications and Pain in Video-assisted Thoracoscopic Surgery Patients Utilizing Continuous Temperature Monitoring
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, The Chief of the department of Anesthesiology, Peking University People's Hospital
Other Study IDs: 2025-h067
Record Dates: First submitted 2025-09-26; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer (Diagnosis); Pain Management; Postoperative Complications; Body Temperature Measurement
MeSH Terms: conditions — Lung Neoplasms; Disease; Agnosia; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Continuous body temperature monitoring — A wireless body temperature transducer is located under the auxiliary. The body temperature is continuously monitored perioperatively.

SUMMARY:
A report from the National Cancer Center (published in JNCC) shows that lung cancer has the highest rates of both new cases and deaths in China. Surgery using a tiny camera (thoracoscopic surgery) is a main treatment for early-stage lung cancer. However, this type of chest surgery carries a much higher risk of patients developing low body temperature during the operation compared to other surgeries. This is because: (1) The surgery is complex and takes longer； (2) The chest cavity is open and exposed to the cool operating room air; (3)General anesthesia affects the brain's ability to regulate temperature and widens blood vessels, causing faster heat loss.Studies show that low body temperature happens in about 65-73% of these chest surgeries, while the average for surgeries longer than 2 hours nationwide is only about 40%.

Low body temperature during surgery isn't just a problem at the time. It also increases the risk of negative outcomes after surgery. As known, it worsens post-surgery pain and increases risks of complications, such as infections, heart problems and bleeding issues.

A common pain control technique for chest surgery is injecting local anesthesia medicine near the spine (Thoracic Paravertebral Block or TPVB). This technique is very effective at reducing pain after surgery, both short-term and long-term. However, new research suggests this nerve block might cause blood vessels to widen, potentially making patients lose body heat faster during surgery. Because TPVB is used so often, it's hard to tell if low body temperature during surgery directly causes worse pain afterwards, or if the nerve block itself influences both temperature and pain. The potential connection between low temperature caused by TPVB and later pain is not yet clear.

The objective of this study is to investigate how low body temperature during and around the time of surgery affects complications after surgery (such as infections, heart and lung problems, longer hospital stays, etc.) in patients undergoing thoracic surgery. The investigators also aim to find the relationship between low body temperature during surgery and the occurrence of pain after surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) I - III
* BMI 18.5 - 30 kg/m²
* Scheduled for Video-assisted thoracoscopic surgery (VATS) lung/mediastinal tumor resection (duration ≥1 hour)
* General anesthesia with regional block (thoracic paravertebral block and serratus anterior plane block)
* Written informed consent.

Exclusion Criteria:

* ASA ≥ IV
* Preoperative fever (>37.5°C) or hypothermia (<36.0°C)
* Chronic pain or opioid use ≥ 3 months
* Immunosuppression
* Thyroid dysfunction
* Neurological dysfunction affecting pain assessment
* Emergency surgery or conversion to thoracotomy
* Planned surgery <1 hour or requiring cardiopulmonary bypass
* Failed regional block (sensory block not covering T2-T8 at 4h postoperation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to accept video-assisted thoracoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | From date of the operation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 days

SECONDARY OUTCOMES:
Pain intensity measured by Numeric Rating Scale on a scale from 0 to 10, where 0 indicates no pain and 10 signifies the worst possible pain. Scores between 1 and 3 typically represent mild pain, 4 to 6 moderate pain, and 7 to 10 severe pain. | From date of the operation until the date of complete remission, assessed up to 30 days
Length of stay | From date of admission to hospital until the date of discharge, assessed up to 30 days
ICU admission rate | From date of the operation until the date of discharge, assessed up to 30 days
30-day readmission rate | From date of discharge until the date of readmission, assessed up to 30 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT07251439/Prot_SAP_000.pdf